CLINICAL TRIAL: NCT04666922
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Rising Intravenous Doses of BI 765080 in Healthy Male Subjects (Single-blind, Randomised, Placebo-controlled, Parallel-group Design)
Brief Title: A Study in Healthy Men to Test How the Body Takes up and Tolerates Different Doses of BI 765080
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1450-0001; 2020-004262-19 (EudraCT Number)
Record Dates: First submitted 2020-12-09; First posted 2020-12-14 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 1 mg BI 765080 (Experimental): BI 765080
  Interventions: Drug: BI 765080
- Placebo group (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo
- 10 mg BI 765080 (Experimental): BI 765080
  Interventions: Drug: BI 765080
- 25 mg BI 765080 (Experimental): BI 765080
  Interventions: Drug: BI 765080
- 50 mg BI 765080 (Experimental): BI 765080
  Interventions: Drug: BI 765080
- 100 mg BI 765080 (Experimental): BI 765080
  Interventions: Drug: BI 765080
- 200 mg BI 765080 (Experimental): BI 765080
  Interventions: Drug: BI 765080

INTERVENTIONS:
Drug: BI 765080 — BI 765080
  Arms: 1 mg BI 765080; 10 mg BI 765080; 100 mg BI 765080; 200 mg BI 765080; 25 mg BI 765080; 50 mg BI 765080
Drug: Placebo — Placebo; 0.9% saline for injection
  Arms: Placebo group

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability, and pharmacokinetics of BI 765080 in healthy male subjects following intravenous administration of single rising doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* A positive poly chain reaction (PCR) test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and clinical symptoms suggestive for this disease on Day -2.
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a Phase I, single-blind, randomized, placebo-controlled, parallel-group design trial to investigate safety, tolerability, and pharmacokinetics of BI 765080 in healthy male subjects following intravenous administration of single rising doses.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 1 mg BI 765080 Group: Subjects received a single dose of 1 milligram (mg) BI 765080 as a 30 minutes (min) intravenous infusion on Day 1.
- 10 mg BI 765080 Group: Subjects received a single dose of 10 milligrams (mg) BI 765080 as a 30 minutes (min) intravenous infusion on Day 1.
- 25 mg BI 765080 Group: Subjects received a single dose of 25 milligrams (mg) BI 765080 as a 30 minutes (min) intravenous infusion on Day 1.
- 50 mg BI 765080 Group: Subjects received a single dose of 50 milligrams (mg) BI 765080 as a 30 minutes (min) intravenous infusion on Day 1.
- 100 mg BI 765080 Group: Subjects received a single dose of 100 milligrams (mg) BI 765080 as a 30 minutes (min) intravenous infusion on Day 1.
- 200 mg BI 765080 Group: Subjects received a single dose of 200 milligrams (mg) BI 765080 as a 30 minutes (min) intravenous infusion on Day 1.
- Placebo Group: Subjects received a single dose of placebo matching BI 765080 as a 30 minutes (min) intravenous infusion on Day 1.
Period: Overall Study
Arm/Group | 1 mg BI 765080 Group | 10 mg BI 765080 Group | 25 mg BI 765080 Group | 50 mg BI 765080 Group | 100 mg BI 765080 Group | 200 mg BI 765080 Group | Placebo Group
Started | 6 | 6 | 6 | 6 | 6 | 6 | 12
Completed | 5 | 6 | 6 | 6 | 6 | 6 | 12
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all subjects who were randomized and treated with at least one dose of study drug. It was used for safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 mg BI 765080 Group | 10 mg BI 765080 Group | 25 mg BI 765080 Group | 50 mg BI 765080 Group | 100 mg BI 765080 Group | 200 mg BI 765080 Group | Placebo Group | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (6.8) | 33.7 (4.0) | 31.2 (7.7) | 38.3 (9.9) | 32.3 (4.9) | 37.5 (11.3) | 32.8 (6.6) | 35.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 5 | 6 | 6 | 12 | 47
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug-related Adverse Events
Description: Percentage of subjects with drug-related adverse events is presented.
Time Frame: Up to 87 days
Population: Treated set (TS): all subjects who were randomised and treated with at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | 1 mg BI 765080 Group | 10 mg BI 765080 Group | 25 mg BI 765080 Group | 50 mg BI 765080 Group | 100 mg BI 765080 Group | 200 mg BI 765080 Group | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Percentage of Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 765080 in Serum Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 765080 in serum over the time interval from 0 extrapolated to infinity (AUC0-∞) is presented.
Time Frame: Within 3 hours (h) prior to administration of BI 765080 and 30 minutes (min), 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h, 72h, 144h, 312h, 480h, 648h, 1320h and 1992h after administration of BI 765080.
Population: Pharmacokinetic parameter analysis set (PKS): all subjects in the treated set (TS) who provided at least one PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability (as specified below). Thus, a subject was included in the PKS, even if he contributed only one PK parameter value for one period to the statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliLitres (h*ng/mL)
Groups:
- 1 mg BI 765080 Group: Subjects received a single dose of 1 milligrams (mg) BI 765080 as a 30 minutes (min) intravenous infusion on Day 1.
Arm/Group | 1 mg BI 765080 Group | 10 mg BI 765080 Group | 25 mg BI 765080 Group | 50 mg BI 765080 Group | 100 mg BI 765080 Group | 200 mg BI 765080 Group
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6
hours*nanograms/milliLitres (h*ng/mL) | 4950 (48.4) | 258000 (20.6) | 973000 (16.2) | 2530000 (39.9) | 7180000 (24.7) | 14900000 (21.8)

3. Secondary Outcome: Maximum Measured Concentration of BI 765080 in Serum (Cmax)
Description: Maximum measured concentration of BI 765080 in serum (Cmax) is presented.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliLitres (ng/mL)
Arm/Group | 1 mg BI 765080 Group | 10 mg BI 765080 Group | 25 mg BI 765080 Group | 50 mg BI 765080 Group | 100 mg BI 765080 Group | 200 mg BI 765080 Group
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6
nanograms/milliLitres (ng/mL) | 274 (21.4) | 3490 (11.0) | 8230 (14.9) | 16900 (29.0) | 35400 (13.7) | 64500 (11.6)

ADVERSE EVENTS:
Time Frame: From first drug administration till end of trial, up to 87 days.
Description: Treated set (TS): all subjects who were randomized and treated with at least one dose of study drug. It was used for safety analyses.
Arm/Group | 1 mg BI 765080 Group | 10 mg BI 765080 Group | 25 mg BI 765080 Group | 50 mg BI 765080 Group | 100 mg BI 765080 Group | 200 mg BI 765080 Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 2/6 | 1/6 | 1/6 | 5/6 | 0/6 | 2/6 | 5/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1 mg BI 765080 Group (N=6) | 10 mg BI 765080 Group (N=6) | 25 mg BI 765080 Group (N=6) | 50 mg BI 765080 Group (N=6) | 100 mg BI 765080 Group (N=6) | 200 mg BI 765080 Group (N=6) | Placebo Group (N=12)
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Reactogenicity event (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT04666922/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT04666922/SAP_001.pdf